CLINICAL TRIAL: NCT02397226
Title: Lower Limb Venous Insufficiency and the Effect of Radiofrequency Treatment Versus Open Surgery. A 5-year Follow-up Using Duplex Ultrasound, Plethysmography, VCSS, AVVQ and EQ-5D
Brief Title: Lower Limb Venous Insufficiency and the Effect of Radiofrequency Treatment Versus Open Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Oskar Nelzén, MD, PhD, University Hospital, Linkoeping
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Varicerstudien
Record Dates: First submitted 2015-03-12; First posted 2015-03-24 (Estimated); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Varicose Veins; Venous Insufficiency
Keywords: Radiofrequency ablation; Plethysmography; Duplex ultrasound; High ligation/stripping
MeSH Terms: conditions — Varicose Veins; Venous Insufficiency | interventions — Radiofrequency Ablation; Conversion to Open Surgery; Catheter Ablation; Anesthesia, General

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Radiofrequency ablation (Active Comparator): Treatment with radiofrequency ablation using radiofrequency ablation catheter. This intervention implies tumescent anesthesia.
  Interventions: Procedure: Radiofrequency ablation; Device: Radiofrequency ablation catheter; Procedure: Tumescent anesthesia
- High ligation/stripping (Active Comparator): Treatment with high ligation/stripping using a vein stripping catheter. This intervention implies general anesthesia.
  Interventions: Procedure: High ligation/stripping; Procedure: General anesthesia; Device: Vein stripping catheter

INTERVENTIONS:
Procedure: Radiofrequency ablation
  Arms: Radiofrequency ablation
Procedure: High ligation/stripping
  Other Names: Open surgery
  Arms: High ligation/stripping
Device: Radiofrequency ablation catheter
  Other Names: Covidien ClosureFast Catheter (7cm)
  Arms: Radiofrequency ablation
Procedure: Tumescent anesthesia
  Arms: Radiofrequency ablation
Procedure: General anesthesia
  Arms: High ligation/stripping
Device: Vein stripping catheter
  Arms: High ligation/stripping

SUMMARY:
200 patients with insufficient great saphenous veins will be randomized to either radiofrequency ablation or high ligation/stripping (open surgery). They will be examined according to standardized examination protocol Venous Clinical Severity Score (VCSS), with duplex ultrasound and plethysmography pre- and postoperatively (1-month, 1-, 3 and 5 years). They are to fill questionnaires EuroQol 5 Dimensions (EQ-5D) and disease specific Aberdeen Varicose Vein Questionnaire (AVVQ).

ELIGIBILITY:
Inclusion Criteria:

* Insufficient great saphenous vein
* Possible to treat with both radiofrequency ablation and high ligation/stripping
* Clinical Etiological Anatomical Pathophysiological score (CEAP) C2-C6

Exclusion Criteria:

* Previous intervention in the affected leg
* Insufficient accessory branch origin close to the great saphenous vein estuary in the femoral vein.
* Small saphenous vein insufficiency with diameter >6 mm and/or flow >100ml/min
* Patient that is not able to perform plethysmography

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2021-11-25 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of treated veins with recanalization using duplex. | 5 years
  Flow detected by duplex at the site of the treated vein.
Number of treated limbs with neovascularization using duplex and/or plethysmography. | 5 years
Prediction of treatment outcome using plethysmography with superficial shut-down. | 1 month postoperatively
  If plethysmography with superficial shut-down of the superficial venous system is able to predict the effect of treatment.

SECONDARY OUTCOMES:
VCSS score | 5 years
  The score of standardized examination protocol VCSS.
AVVQ score | 5 years
  The score of disease specific questionnaire AVVQ
EQ-5D score | 5 years
  The score of EQ-5D questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Helene Zachrisson, Associate Professor, MD, Study Chair — Linkoeping University; Oskar Nelzén, MD, Principal Investigator — Linkoeping University
Locations (2):
- Sweden (2):
  - University Hospital Linköping, Linköping, Östergötland County
  - Vrinnevisjukhuset, Norrköping, Östergötland County

REFERENCES:
- [Derived] Nelzen POE, Skoog J, Oster M, Zachrisson H. Impact on venous haemodynamics after treatment of great saphenous vein incompetence using plethysmography and duplex ultrasound. Phlebology. 2020 Aug;35(7):495-504. doi: 10.1177/0268355519898952. Epub 2020 Jan 20. PMID 31959059